CLINICAL TRIAL: NCT06981715
Title: Investigation of the Efficacy of Extracorporeal Shock Wave Therapy and Kinesiotaping Applied as an Addition to Conservative Treatment in Individuals With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758!
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel syndrome; treatment; kinesiotaping
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): Control Group:
  Resting splint fixing the ankle in neutral position
  Worn every night before going to bed, used for 6-8 hours
  Objective: To reduce the pressure on the median nerve
  Exercise Programme:
  Applied 1-2 times a day
  Each exercise 10 repetitions, 2 sets
  Content:
  Nerve mobilisation exercises (median nerve sliding and stretching)
  Wrist stretching and flexor-extensor tendon sliding exercises
  Finger opening-closing, fist making exercises
  Interventions: Other: Conservative treatment
- ESWT group (Experimental): ESWT group:
  Resting splint fixing the ankle in neutral position
  Worn every night before going to bed, used for 6-8 hours
  Objective: To reduce the pressure on the median nerve
  Exercise Programme:
  Applied 1 time per day
  Each exercise 10 repetitions, 2 sets
  Content:
  Nerve mobilisation exercises (median nerve sliding and stretching)
  Wrist stretching and flexor-extensor tendon sliding exercises
  Finger opening-closing, fist making exercises
  ESWT Protocol:
  Device Radial ESWT device
  Area of application Wrist volar surface (carpal tunnel area)
  Parameters
  Frequency: 5 Hz
  4 Bar
  Number of beats 2000 pulses/session
  Application time 5-10 minutes per session
  Interventions: Other: Conservative treatment; Other: ESWT
- ESWT+Taping Group (Experimental): ESWT+Taping Group:
  Resting splint fixing the ankle in neutral position Worn every night before going to bed, used for 6-8 hours Objective: To reduce the pressure on the median nerve
  Exercise Programme:
  Applied 1 time per day Each exercise 10 repetitions, 2 sets
  Content:
  Nerve mobilisation exercises (median nerve sliding and stretching) Wrist stretching and flexor-extensor tendon sliding exercises Finger opening-closing, fist making exercises
  ESWT Protocol:
  Device Radial ESWT device Area of application Wrist volar surface (carpal tunnel area) Parameters Frequency: 5 Hz 4 Bar Number of beats 2000 pulses/session
  Kinesiobanding technique Kinesio taping was performed with the Button hole technique described by Dr Kenzo Kase. In this technique, a kinesio tape was measured and cut from the medial and lateral epicondyle level on the palmar side of the forearm, from the base of the proximal phalanges to the epicondyles of the humerus on the dorsal side of the forearm.
  Interventions: Other: Conservative treatment; Other: ESWT; Other: Kinesiotaping

INTERVENTIONS:
Other: Conservative treatment — Night Splint Resting splint fixing the ankle in neutral position
  Worn every night before going to bed, used for 6-8 hours
  Objective: To reduce the pressure on the median nerve
  Exercise Programme:
  Applied 1-2 times a day
  Each exercise 10 repetitions, 2 sets
  Content:
  Nerve mobilisation exercises (median nerve sliding and stretching)
  Wrist stretching and flexor-extensor tendon sliding exercises
  Finger opening-closing, fist making exercises
Other: ESWT — ESWT Protocol:
  Device Radial ESWT device Area of application Wrist volar surface (carpal tunnel area) Parameters Frequency: 5 Hz 4 Bar Number of beats 2000 pulses/session Application time 5-10 minutes per session
  Arms: ESWT group; ESWT+Taping Group
Other: Kinesiotaping — Kinesio taping was performed with the Button hole technique described by Dr Kenzo Kase. In this technique, a kinesio tape was measured and cut from the medial and lateral epicondyle level on the palmar side of the forearm, from the base of the proximal phalanges to the epicondyles of the humerus on the dorsal side of the forearm. The tape was folded and the midpoint was found, 2 short incisions were made and 2 button holes were obtained through which the 3rd and 4th finger would pass. The paper behind the band was torn and the 3rd and 4th fingers were passed through the holes. The patient's wrist was brought to extension and radial deviation and the tape was glued with a slight (15-25%) tension towards the medial epicondyle on the palmar side of the forearm. Then the wrist was flexed and ulnar deviated and the tape was glued with a slight (15-25%) tension towards the lateral epicondyle.
  Arms: ESWT+Taping Group

SUMMARY:
This study was conducted to compare the effectiveness of different treatment combinations in individuals with carpal tunnel syndrome (CTS). Participants were divided into three groups: The control group received only night splinting and exercise programme, while the second group received extracorporeal shock wave therapy (ESWT) in addition. The third group received kinesiobanding in addition to night splinting, exercise and ESWT. The study evaluates the effect of multimodal conservative treatment approaches on CTS symptoms and aims to demonstrate the additional benefits of ESWT and kinesiobanding in particular. The findings provide important clues for clinical practice.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common entrapment neuropathy resulting from compression of the median nerve at the wrist level, with symptoms such as paresthesia, pain and loss of muscle strength. This study comparatively evaluated the effects of different conservative treatment combinations on symptoms and functional status in individuals with CTS. Participants were divided into three groups. The control group received the standard conservative approach of night splinting and exercise programme. Extracorporeal shock wave therapy (ESWT) group received ESWT, which is known to increase tissue regeneration and blood flow, in addition to night splinting and exercise. In the ESWT+Taping group, in addition to night splinting, exercise and ESWT, kinesiobanding, which aims to provide proprioceptive support and reduce oedema, was applied. Pain intensity, symptom severity, functionality, hand grip strength and electrophysiological parameters were evaluated before and after treatment. This study draws attention to the importance of multidisciplinary and holistic approaches in the treatment of CTS and offers important contributions to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 who applied to Ahi Evran University Physical Medicine and Rehabilitation Outpatient Clinic and were diagnosed with moderate or mild carpal tunnel syndrome by clinical, physical examination and EMG
* Patients who understand and can apply the patient information form
* Patients who gave consent and participated in the study according to the informed consent form

Exclusion Criteria:

* Cervical radiculopathy
* Polyneuropathy
* Brachial plexopathy
* History of trauma or fracture of the wrist and forearm
* Systemic corticosteroid use, history of malignancy
* History of carpal tunnel syndrome surgery
* Pregnant and lactating women
* Severe carpal tunnel syndrome, tenar atrophy on physical examination 9.
* Patient reluctance to participate in treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-05-17 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 5 week
  Visual Analogue Scale (VAS) was used to determine the presence and severity of low back pain in the study participants. GAS is a practical test with high validity and reliability in pain assessment. GAS is an assessment method numbered from 0 to 10, where '0' indicates no pain and '10' indicates the presence of the most severe pain. Participants were asked to mark the degree of pain they had on this scale and recorded.

SECONDARY OUTCOMES:
Symptom Severity and Functionality | 5 week
  It was developed by Levine et al. in 1993 (102). In 2006, its Turkish validity and reliability was performed by Sezgin et al. This scale used for clinical standardisation of CTS consists of nineteen questions. The answers vary between one and five points. A high mean score indicates that the patient has low functional capacity and severe symptoms. The questionnaire consists of two parts, the Boston Symptom Severity Scale (SSS) and the Boston Functional Status Scale (FSS). The Boston-SSS has 11 questions and responses range from 'none (1 point)' to 'very severe (5 points)'. The Boston-FDS has 8 questions and the answers range from 'very easy (1 point)' to 'very difficult (5 points)'. The patient's score is divided by the total score and a ratio between 0 and 1 is obtained. A ratio closer to 1 indicates an increase in dysfunction and symptom severity.
Hand Grip Strength | 5 week
  The Jamar dynamometer was used to measure gross grip strength. Jamar dynamometer measures static grip strength in kilograms. The measurements were performed in the position recommended by the American Society of Hand Therapists, with the patient sitting, arm in adduction, elbow flexed 90 degrees, forearm in neutral position. Patients were asked to squeeze the dynamometer with maximum strength for at least 3 seconds. 3 measurements were made and the measurements were made at 1 minute intervals and the mean was recorded in kilograms.
Electrophysiological Assessments | 5 week
  A Nihon Kohden Neuropack S1 MEB-9400 electroneuromyography (ENMG) device (Nihon Kohden Corp., Tokyo, Japan) was utilized. Values of median sensory distal latency (mSDL) <3.6 ms, and median sensory nerve conduction velocity (mSNCV) >50 m/s were deemed normal. The classification for CTS provided by the American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) was utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, PhD., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No